CLINICAL TRIAL: NCT04778046
Title: Defining a Noninvasive Signature for Pulmonary Vascular Remodeling in Group 3 PH
Brief Title: Pulmonary Hypertension SOLAR
Acronym: PH SOLAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Associate Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00106221
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-01

CONDITIONS: Interstitial Lung Disease; COPD; Pulmonary Arterial Hypertension
Keywords: Lung Transplant; Group 3 PH
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- PAH: (Experimental): Clinical diagnosis of PAH (Group 1 PH) in the absence of severe chronic lung disease, left heart disease, chronic thromboembolism, sarcoidosis, sickle cell disease or other causes of non-Group 1 PH.
  Interventions: Drug: Hyperpolarized 129Xe
- COPD-noPH (Experimental): Clinical diagnosis of COPD in the absence of precapillary PH.
  Interventions: Drug: Hyperpolarized 129Xe
- COPD-PH (Experimental): Clinical diagnosis of COPD with precapillary PH
  Interventions: Drug: Hyperpolarized 129Xe
- IPF-noPH (Experimental): Clinical diagnosis of IPF in the absence of precapillary PH
  Interventions: Drug: Hyperpolarized 129Xe
- IPF-PH (Experimental): Clinical diagnosis of IPF with precapillary PH
  Interventions: Drug: Hyperpolarized 129Xe

INTERVENTIONS:
Drug: Hyperpolarized 129Xe — Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC),
  Other Names: Xe MRI

SUMMARY:
The main goal of this study is to develop a noninvasive signature for pulmonary vascular remodeling in Group 3 PH patients, using hyperpolarized 129Xe magnetic resonance imaging (129Xe MRI). Such a signature may identify Group 3 PH responders to PAH-specific therapies. PAH's unique 129Xe MRI signature has been shown in previous studies. Past studies have lacked a pathologic "ground truth" correlate of these signatures, which could be provided by comparing them with the pathology of lung explant tissue from patients who have undergone a lung transplant. This signature could be validated in a cohort of patients with Group 3 PH in future studies.

DETAILED DESCRIPTION:
The objective of this study is to identify a 129Xe MRI signature associated with PAH-like pulmonary vascular remodeling, consisting of plexiform arteriopathy, smooth muscle cell proliferation, and vascular fibrosis, in IPF and COPD that could be used to identify potential responders vs non-responders to PAH-specific therapies. The central hypothesis is that similar mechanisms and pathways underlie pulmonary vascular remodeling in IPF-PH, COPD-PH, and PAH. However, only a subset of Group 3 PH patients display remodeling consistent with PAH, resulting in responder vs. non-responder phenotypes when treated with PAH-specific therapies. In preliminary studies of subjects treated with Tyvaso, The study team has observed distinct 129Xe MRI signatures at baseline and with therapy depending on patients' underlying lung function. Consistent with this, recent studies using single-cell RNA sequencing (scRNAseq) of the pulmonary vasculature in IPF have demonstrated changes consistent with vascular remodeling.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years' old
2. Be on the lung transplant waiting list at Duke University Medical Center.
3. PH as defined by RHC - mPAP > 20 mmHg, PVR > 3 WU, PCWP < 15 mmHg
4. Groups defined as:

   PAH: Clinical diagnosis of PAH (Group 1 PH) in the absence of severe chronic lung disease, left heart disease, chronic thromboembolism, sarcoidosis, sickle cell disease, or other causes of non-Group 1 PH.

   COPD-noPH: Clinical diagnosis of COPD in the absence of precapillary PH.

   COPD-PH: Clinical diagnosis of COPD with precapillary PH.

   IPF-noPH: Clinical diagnosis of IPF in the absence of precapillary PH.

   IPF-PH: Clinical diagnosis of IPF with precapillary PH.
5. Willing and able to give informed consent and adhere to visit/protocol schedules (consent must be given before any study procedures are performed).

Exclusion Criteria:

1. Moderate to severe heart disease (LVEF < 45% or severe LV Hypertrophy).
2. Sarcoidosis.
3. Active cancer.
4. Sickle cell anemia.
5. Liver disease (Childs-Pugh class C).
6. Prisoners and pregnant women will not be approached for the study.
7. Inability to obtain consent.
8. Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine).
9. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
a pathology-based 129Xe MRI noninvasive signature of pulmonary vascular remodeling that could be validated in a larger cohort of Group 3 PH patients | Day 1
  Such a signature could then be tested in clinical trials in Group 3 PH. These studies will have an important positive impact because they lay the foundation for a precision medicine strategy in Group 3 PH through the identification of potential responders and non-responders to PAH-specific therapies

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Rajagopal, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No